CLINICAL TRIAL: NCT07240649
Title: Emerging Indications for Hyperbaric Oxygen Treatment
Brief Title: Outcomes From Hyperbaric Oxygen (HBO2) Treatment for Emerging Indications
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jay C. Buckey Jr. (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Sponsor-Investigator, Jay C. Buckey Jr., Principal Investigator, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02003096
Record Dates: First submitted 2025-10-26; First posted 2025-11-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Post-COVID-19 Condition; Ulcerative Colitis; Crohn Disease; Calciphylaxis; Frostbite; Acute COVID-19; Pyoderma Gangrenosum; Pterygium; Hypospadias; Head Trauma; Pneumatosis Intestinalis; Ischemic Bowel; Raynaud Syndrome; Malignant Otitis Externa; Nonarteritic Anterior Ischemic Optic Neuropathy; Central Retinal Vein Occlusion; Femoral Head Necrosis; Invasive Fungal Infection; Chronic Anal Fissure; Vasculitic Ulcer; Graft-vs-Host Disease; Decubitus Ulcer; Greater Trochanteric Pain Syndrome; Rectovaginal Fistula; Pouchitis; Tinnitus; Clostridium Enterocolitis; Branch Retinal Artery Occlusion; Axonotmesis; Multiple Sclerosis; Inclusion Body Myositis; Epidermolysis Bullosa (EB); Osteonecrosis; Ulcer Ischemic; Avascular Necrosis of Bone; Prosthesis Related Infections; Facial Filler Injections; Cystitis Chronic; Ligament Injury; Anastomosis, Leaking; Cartilage Injury
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Calciphylaxis; Frostbite; Pyoderma Gangrenosum; Pterygium; Hypospadias; Craniocerebral Trauma; Raynaud Disease; Optic Neuropathy, Ischemic; Retinal Vein Occlusion; Invasive Fungal Infections; Graft vs Host Disease; Pressure Ulcer; Rectovaginal Fistula; Pouchitis; Tinnitus; Enterocolitis, Pseudomembranous; Retinal Artery Occlusion; Trauma, Nervous System; Multiple Sclerosis; Myositis, Inclusion Body; Epidermolysis Bullosa; Osteonecrosis; Prosthesis-Related Infections | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hyperbaric oxygen treated group (Experimental): This individuals will be receiving hyperbaric oxygen treatment for the condition listed in the conditions section. Patients come daily for the treatment and receive hyperbaric oxygen at 2.0-2.4 atmospheres absolute for 90 minutes at the treatment pressure.
  Interventions: Device: Hyperbaric oxygen treatment (HBOT); Drug: 100% Oxygen

INTERVENTIONS:
Device: Hyperbaric oxygen treatment (HBOT) — Hyperbaric oxygen refers to oxygen given at pressures higher than atmospheric pressure (higher than 1.4 ATA) in pressurized chamber.
  Other Names: HBO2
Drug: 100% Oxygen — Receiving 100% oxygen as part of HBOT
  Other Names: O2

SUMMARY:
This study will evaluate the effectiveness of hyperbaric oxygen therapy (HBOT) on treating emerging indications (i.e., conditions that have shown to potentially benefit from HBOT) using the Multicenter Registry for Hyperbaric Oxygen Treatment. The study team aims to collect ongoing data on how well HBOT treats these emerging indications, and to add these data to the growing HBO Registry. The research team hypothesizes that HBOT will result in improvements of the condition of the various emerging indications.

DETAILED DESCRIPTION:
Currently, the Undersea and Hyperbaric Medical Society (UHMS) has identified 15 conditions where HBO2 can be considered an approved treatment. These range from decompression illness, where the combination of increased pressure, relief of hypoxia, and reduced inflammation from HBO2 help combat the impaired circulation and endothelial damage caused by bubbles, to radiation injury, where the pulses of oxygen promote angiogenesis and wound healing. Because of HBO2's effects on hypoxia and inflammation, more medical diagnoses exist that can benefit from HBO2. HBO2 is typically given in long courses (20-40 treatments), however, and most centers see only a limited number of patients. Therefore, gathering outcome data on HBO2 treatment has been limited, and often, only case reports or small case series are available to support its use. In addition, practice patterns differ across centers, and some centers may use HBO2 successfully for an indication that other centers may not consider it for. To gather more data on HBO2 applications, outcome data from multiple centers need to be combined. The goal of the Multicenter Registry for Hyperbaric Oxygen Treatment is to collect and aggregate these data.

In a recent publication from our group, we presented data for 45 emerging indications for hyperbaric oxygen treatment. A unifying theme among many of these indications is that they involve hypoxia and/or inflammation as prime drivers of the pathology.

For many of the indications the use of HBOT is based on the underlying pathophysiology, where the presence of hypoxia and/or inflammation indicates that HBOT might be useful. The outcome data, however, are based on case reports or small case series. This project will collect consistently acquired outcome data for indications where HBOT is being used, but the underlying data supporting its use is limited.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for HBOT with an emerging indication

Exclusion Criteria:

* Contraindication to hyperbaric oxygen treatment (untreated seizures, pneumothorax, significant pulmonary airspace pathology that might lead to pulmonary barotrauma, unmanageable confinement anxiety, chronic obstructive pulmonary disease with CO2 retention)
* Pregnant persons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Life EuroQOL EQ-5D-5L Questionnaire | Within one week of starting HBO2 and within one week of ending HBO2 treatment
  Every individual has quality of life measured using the EuroQol EQ-5D-5L measure. The measure has 5 scales (Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression), that each have 5 levels (none, slight, moderate, severe, unable). The scores are calculated using the procedures outlined in the EuroQOL handbook to create a final score on a 0-1 scale. There is also an overall visual analog scale that asks about perceived health on a 0-100 scale. Higher scores indicate better quality of life. Data are aggregated in the Multicenter Registry for Hyperbaric Oxygen Treatment.

SECONDARY OUTCOMES:
Urogenital Distress Inventory | Within one week of starting HBO2 treatments and within one week completing HBO2 treatments
  Patients with cystitis will complete the Urinogential Distress Inventory (UDI). The six questions ask about symptoms on a 4 point scale (No= 0, Not at all= 1, Somewhat= 2, Moderately= 3, Quite a bit= 4). The UDI scaled score is calculated by adding all scores and multiplying by 6 and then multiply by 25 for the scale score. Missing items are dealt with by using the mean from the answered items only. Higher score = higher disability.
Bowel symptoms questionnaire | Within one week of starting HBO2 treatments and within one week completing HBO2 treatments
  Those with conditions affecting the gastrointestinal tract will complete the bowel symptoms questionnaire. The questionnaire has nine questions that cover the areas of frequency, blood, pain, and urgency. Severity is rated on a 4 point scale from 0 to 4 with 4 being severe. Higher values indicate more symptoms.
Head and Neck Questionnaire | Within one week of starting HBO2 treatments and within one week completing HBO2 treatments
  The head and neck questionnaire has 37 questions selected from the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-H&N35 and the Groningen Radiotherapy-Induced Xerostomia (GRIX) questionnaire. The questionnaire covers dry mouth, pain, and difficulties with smell and taste. The scores are converted to a 0-100 scale with higher numbers indicating more symptoms.
Perianal Crohn's Symptom Index Questionnaire | Within one week of starting HBO2 treatments and within one week completing HBO2 treatments
  The perianal Crohn's symptom index has 13 questions that cover fistulas, fistula discharge, rectal discharge, bowel frequency, urgency, blood, and pain. The answers are converted to an overall summed score with higher levels indicating more symptoms.
Hip dysfunction and Osteoarthritis Outcome Score (HOOS) Questionnaire | Within one week of starting HBO2 treatments and within one week completing HBO2 treatments
  Individuals with conditions involving the knee or hip will complete the HOOS questionnaire. The questions are divided into symptoms, stiffness, pain, function (daily living), function (sports), and quality of life. Symptoms are measured on a 5 point scale from none to extreme. The answers are computed into individual sub scales for each major area and an overall total score. Higher numbers indicate more symptoms.
Wound Score (Strauss Score) | Within one week of starting HBO2 treatments and within one week completing HBO2 treatments
  Individuals with wounds will have the wound (Strauss) score completed. The score covers five areas (Appearance, Size, Depth, Infection/Bioburden, and Perfusion). Each area is graded from best (2 points) to worst (0 points). Depth also has a possible 1.5 score for subcutaneous tissue involvement. Higher scores are better with healthy wounds in the 7.5 to 10 point range.
Subjective Assessment | Within one week of starting HBO2 treatments and within one week completing HBO2 treatments
  For all enrollees a 4 level subjective assessment will be completed. The scale ranges from 1 resolved/healed to 4 worse with higher levels indicating less improvement.
Calciphylaxis Measurement Package | Within one week of starting HBO2 treatments and within one week completing HBO2 treatments
  For individuals treated for calciphylaxis, data will be collected on the following parameters:
  Number of wounds Pre and post wound measurements in cm Number of surgical interventions
Frostbite Measurement Package | Within one week of starting HBO2 treatments and within one week completing HBO2 treatments
  For all individuals treated for frostbite data will be collected on:
  Number of wounds Wound measurements in cm Number of surgical interventions
Pyoderma Gangrenosum Measurement Package | Within one week of starting HBO2 treatments and within one week completing HBO2 treatments
  For all individuals treated for pyoderma gangrenous data will be collected on:
  Number of wounds Wound measurements in cm Number of surgical interventions
Raynaud Syndrome Measurement Package | Within one week of starting HBO2 treatments and within one week completing HBO2 treatments
  For all individuals treated for Raynaud's data will be collected on:
  Number of wounds Wound measurements in cm Number of surgical interventions

CONTACTS AND LOCATIONS:
Overall Officials: Jay Buckey, Principal Investigator — Dartmouth-Hichcock Medical Center

REFERENCES:
- [Background] Tanaka HL, Rees JR, Zhang Z, Ptak JA, Hannigan PM, Silverman EM, Peacock JL, Buckey JC; Multicenter Registry for Hyperbaric Oxygen Treatment Consortium. Emerging Indications for Hyperbaric Oxygen Treatment: Registry Cohort Study. Interact J Med Res. 2024 Aug 20;13:e53821. doi: 10.2196/53821. PMID 39078624
- [Background] Harlan NP, Ptak JA, Rees JR, Cowan DR, Fellows AM, Moses RA, Kertis JA, Hannigan PM, Juggan SA, Peacock J, Bennett M, Buckey JC. International Multicenter Registry for Hyperbaric Oxygen Therapy: Results through June 2021. Undersea Hyperb Med. 2022 Third Quarter;49(3):275-287. PMID 36001560
- [Background] Harlan NP, Ptak JA, Rees JR, Cowan DR, Fellows AM, Kertis JA, Hannigan PM, Peacock JL, Buckey JC. Development of an International, Multicenter, Hyperbaric Oxygen Treatment Registry and Research Consortium: Protocol for Outcome Data Collection and Analysis. JMIR Res Protoc. 2020 Aug 17;9(8):e18857. doi: 10.2196/18857. PMID 32579537
- [Background] 1. Huang ET. Hyperbaric Medicine Indications Manual. 15th ed. North Palm Beach, FL: Best Publishing Company; 2023 2023. 445 p.